CLINICAL TRIAL: NCT05031351
Title: Nuclear Factor Kappa Beta Inhibition in Patients With Amyotrophic Lateral Sclerosis: A Phase II Randomized Placebo Controlled Trial
Brief Title: NF-κB Inhibition in Amyotrophic Lateral Sclerosis
Acronym: NIALS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 032-2017
Record Dates: First submitted 2021-08-05; First posted 2021-09-01 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: ALS
Keywords: Withania somnifera; Ashwagandha; Nuclear Factor Kappa Beta Inhibition; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dosage Withania somnifera (Experimental): 544mg oral twice a day
  Interventions: Drug: Withania somnifera
- Medium dosage Withania somnifera (Experimental): 272mg oral twice a day
  Interventions: Drug: Withania somnifera
- Placebo (Placebo Comparator): Matched capsules twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Withania somnifera — Nuclear Factor Kappa Beta Inhibitor
  Arms: High dosage Withania somnifera; Medium dosage Withania somnifera
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This is a Phase II, single centre, randomized, parallel, double blind, placebo-controlled clinical trial to determine the safety of Withania somnifera in participants with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
There will be up to 75 participants randomized 1:1:1 to receive either high dosage Withania somnifera extract (1088 mg daily), medium dosage Withania somnifera extract (544 mg daily) or matching placebo. The study will consist of a Screening Period, Randomization visit, Baseline visit, and Follow-up visits. The treatment period will be 8 weeks and a final follow up call will occur at Week 9.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with laboratory supported probable, clinically possible, probable or definite ALS according to the World Federation of Neurology Revised El Escorial criteria (83) (Appendix A)
* Disease duration from symptom onset no greater than 36 months at the Screening Visit
* Aged 18 years or older
* Capable of providing informed consent and complying with study procedures
* If taking riluzole, on a stable dose for at least 30 days prior to Screening Visit
* If taking edaravone, on a stable dose for at least one cycle prior to Screening Visit
* If on BiPAP, average usage of no more than 12 hours per day at time of Screening Visit
* Able to swallow a capsule at Baseline Visit
* Fluency in English or French

Exclusion Criteria:

* Exposure to any investigational agent or Withania somnifera (Ashwagandha) within 30 days prior to the Screening Visit; simultaneous participation in other observational studies is allowed upon Site Investigator approval
* Presence of any of the following clinical conditions:

  1. Substance abuse within the past year
  2. Unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active malignancy or infectious disease
  3. Acquired Immunodeficiency Syndrome (AIDS) or AIDS-related complex
  4. Unstable psychiatric illness defined as psychosis (hallucinations or delusions) or untreated major depression within 90 days prior to the Screening Visit
* Hypersensitivity or allergy to Withania somnifera
* Uncontrolled diabetes with severe associated complications (such as neuropathy)
* Untreated hypertension, active stomach ulcers, or untreated thyroid disorder
* Previously diagnosed auto-immune condition with or without neurological manifestations (e.g. multiple sclerosis (MS), systemic lupus erythematosus (SLE), rheumatoid arthritis, etc.)
* Current or planned use of oral, intramuscular or intravenous steroid drugs (such as prednisone, prednisolone, dexamethasone, triamcinolone, methylprednisolone, oxandrolone, and others) or immunosuppressant drugs (azathioprine, mycophenolate, tacrolimus, sirolimus, cyclophosphamide, and others) for more than 7 days
* Planned consumption of alcohol, other drugs or natural health products with sedative and anxiolytics properties while taking study drugs (8 week duration)
* Current or planned use of continuous subcutaneous, intravenous or oral anticoagulant drugs
* Scheduled for surgery under general anesthetic within 14 days of Screening Visit
* Pregnancy or planned pregnancy. Women of childbearing potential must have a negative pregnancy test and be non-lactating at the Screening Visit
* Insertion of a diaphragm pacing system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (safety) | From Baseline visit until end of study visit (Week 9)
  Incidence of adverse events

SECONDARY OUTCOMES:
Change in SICI values | Baseline to 8 weeks
  Short-interval intracortical inhibition (SICI) measured by transcranial magnetic stimulation (TMS).
Change in RMT values | Baseline to 8 weeks
  Resting motor threshold (RMT) measured by transcranial magnetic stimulation (TMS).
Change in recovery cycle | Baseline to 8 weeks
  This is a lower motor neuron excitability parameter measured by threshold tracking nerve excitability testing (NET).
Change in strength duration time constant | Baseline to 8 weeks
  This is a lower motor neuron excitability parameter measured by threshold tracking nerve excitability testing (NET).

OTHER OUTCOMES:
Incident cases of ALSFRS-R score changes of 4 or more points | Baseline to 9 weeks
  Any incident case of ≥ 4-point increase in the ALS Functional Rating Scale-Revised (ALSFRS-R) scores or significant clinical improvement at week 8 will be reported. Changes in pro-inflammatory tests (CRP and IL-6) from baseline to Week 8 will be assessed.
Change in serum IL-6 levels | Baseline to 8 weeks
  Serum IL-6 levels will serve as an indirect marker of NF-kB inhibition and target engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Agessandro Abrahao, MD, MSc, Principal Investigator — Sunnybrook Research Institute, University of Toronto; Lorne Zinman, MD, MSc, Study Director — Sunnybrook Research Institute, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada